CLINICAL TRIAL: NCT04368624
Title: A Novel Approach Integrating Non-invasive Skin Tape-stripping to Evaluate and Monitor Patients With Phenylketonuria (PKU)
Brief Title: PKU Skin Stripping
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-3664
Record Dates: First submitted 2020-04-15; First posted 2020-04-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — Surgical Tape; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PKU: 1. Patients with classical PKU phenotype (serum phenylalanine concentration > 10 mg/dL on a normal diet at diagnosis) # ~25
  2. Patients with hyperphenylalaninemia (serum phenylalanine concentration < 10 mg/dL on a normal diet at diagnosis) # ~15
  3. Patients with PKU on therapy with Kuvan # ~10
  Interventions: Other: Skin Tape; Diagnostic Test: Blood Draw
- Non-PKU Control: Study Controls: Up to 50 children and adults without a known metabolic disorder.
  Interventions: Other: Skin Tape

INTERVENTIONS:
Other: Skin Tape — Skin sample collection: samples of human stratum corneum will be obtained with squame adhesive tape disks typically at the time of their clinic appointment. The tape will be placed on the inside of the forearm and the procedure will be repeated up to five times per patient to have sufficient corneocytes for analysis. This type of sampling is non-invasive.
Diagnostic Test: Blood Draw — Blood specimens: blood will be obtained for serum amino acids/phenylalanine levels. This sample is obtained for disease monitoring as part of routine standard of care. Results from up to three clinic visits will be correlated with the tape sample obtained on the same day.
  Groups: Participants with PKU

SUMMARY:
PURPOSE OF STUDY: To determine if a non-invasive skin stripping technique can be used to detect individuals with phenylalanine abnormalities, and to monitor dietary and/or drug effects over time.

DETAILED DESCRIPTION:
This study will determine if a non-invasive skin stripping technique can be used to detect individuals with phenylalanine abnormalities, and to monitor dietary and/or drug effects over time. To do this 50 children and adults with phenylalanine abnormalities and up to 50 unaffected controls will be recruited to this study. The 50 affected individuals will have their metabolomic profile analyzed from up to 3 skin-stripping samples over time and compared to their serum amino acid profile in both dried blood spots and a typical blood sample. The unaffected controls will provide one skin-stripping sample. Clinical data regarding compliance with dietary therapy and other medications will be collected to determine other effects on the metabolome.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of PKU that is confirmed by elevated serum phenylalanine.
2. Any age.
3. Subject or the subject's legal authorized representative has given written informed consent to participate in the study.

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Phenylketonuria (PKU) is a serious metabolic disorder characterized by intolerance to the dietary intake of phenylalanine. When untreated, older children can show the following clinical manifestations: microcephaly, epilepsy, a musty body odor, decreased skin and hair pigmentation, eczema, severe intellectual disability, and behavioral problems.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Control Metabolomic Profile (skin) | 5 years
  The establishment of normative data for the skin metabolome will provide a baseline for assessing changes in the skin metabolome that occur during development and with disease.
  By exhaustive extraction of the adhesive tapes with organic solvents, the investigators will analyze the metabolome of the stratum corneum with developed targeted methods for amino acids. The analysis will be performed using ultra high performance liquid chromatography - quadrupole time of flight mass spectrometry (UPLCQTOF-MS) to identify biochemical changes in the tape-stripped skin metabolome. With the comparative intensity/concentration results of identified metabolites, a subsequent metabolic network reconstruction will be carried out to reveal the underlying mechanism perturbed in PKU and metabolic response to diet or therapeutic interventions.
PKU Metabolomic Profile (skin) | 5 years
  By exhaustive extraction of the adhesive tapes with organic solvents, the investigators will analyze the metabolome of the stratum corneum with developed targeted methods for amino acids. The analysis will be performed using ultra high performance liquid chromatography - quadrupole time of flight mass spectrometry (UPLCQTOF-MS) to identify biochemical changes in the tape-stripped skin metabolome. With the comparative intensity/concentration results of identified metabolites, a subsequent metabolic network reconstruction will be carried out to reveal the underlying mechanism perturbed in PKU and metabolic response to diet or therapeutic interventions.
Metabolomic Profile Change | 5 years
  Determine if the metabolomic profile changes over time in patients with PKU. By exhaustive extraction of the adhesive tapes with organic solvents, the investigators will analyze the metabolome of the stratum corneum with developed targeted methods for amino acids. The analysis will be performed using ultra high performance liquid chromatography - quadrupole time of flight mass spectrometry (UPLCQTOF-MS) to identify biochemical changes in the tape-stripped skin metabolome. With the comparative intensity/concentration results of identified metabolites, a subsequent metabolic network reconstruction will be carried out to reveal the underlying mechanism perturbed in PKU and metabolic response to diet or therapeutic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Prada, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holleran WM, Ziegler SG, Goker-Alpan O, Eblan MJ, Elias PM, Schiffmann R, Sidransky E. Skin abnormalities as an early predictor of neurologic outcome in Gaucher disease. Clin Genet. 2006 Apr;69(4):355-7. doi: 10.1111/j.1399-0004.2006.00589.x. No abstract available. PMID 16630170